CLINICAL TRIAL: NCT06124261
Title: Androgens and Nonalcoholic Fatty Liver Disease (NAFLD) In Reproductive-Aged Women With and Without Polycystic Ovary Syndrome (PCOS)
Brief Title: Androgens and NAFLD Longitudinal Cohort Study
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Duke University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-39040; 1R01DK134633-01A1 (NIH)
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: PCOS; NAFLD; NASH
Keywords: Androgen
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood samples and optional liver samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MASLD and PCOS hyperandrogenism: Patients with MASLD and PCOS with the phenotype of hyperandrogenism
- MASLD and PCOS non-hyperandrogenism: Patients with MASLD and PCOS with the phenotype of non-hyperandrogenism
- MASLD and no-PCOS: Patients with metabolic dysfunction-associated steatotic liver disease (MASLD) and no PCOS

SUMMARY:
The researchers want to learn how androgens, a type of sex hormone, might affect nonalcoholic fatty liver (NAFLD) in young women over time. NAFLD happens when fat builds up in the liver which can cause damage to the liver such as inflammation or scarring.

Young women with a condition called polycystic ovary syndrome (PCOS) have a high risk for NAFLD, and they often have high androgen levels too. So the researchers are recruiting young women with PCOS as well as those without PCOS, and will compare changes in NAFLD over time between young women with and without PCOS.

This study is funded by the National Institutes of Health

DETAILED DESCRIPTION:
The studies central hypothesis is that androgens promote liver injury and NAFLD/NASH progression in PCOS, which occurs through aberrant lipid activity (including lipotoxicity and dysregulated de novo lipogenesis), in part from androgenic effects on visceral adipose tissue (VAT). Data in young women taking exogenous testosterone show redistribution of fat from subcutaneous to visceral stores In the general population, VAT promotes NASH through several established pathways, including production of tissue injurious or "lipotoxic" lipids such as some phospholipid, sphingomyelin, and ceramide species. Recent data show androgen- associated increase in serum glycerophospholipids in women with PCOS, a lipid class that is associated with NASH in women. Additionally, androgen-associated de novo lipogenesis (DNL) may contribute to NASH in women. Hepatic DNL is a key source of lipid accumulation, and co-investigators at Duke University recently discovered an enzymatic balance that regulates hepatic DNL with dysregulation of this pathway (reflected by branched-chain keto and amino acids) predictive of prevalent NASH in humans. Androgen-induced de novo lipogenesis also occurs in cultured hepatocytes from women (but not men) supporting the researchers focused evaluation of the relationship between androgens, dysregulated hepatic DNL, and NASH in PCOS.

As existing data support androgenic effects on hepatic and visceral fat in women, the researchers will now determine the relationship of androgens with liver injury and progression in PCOS and the potential mechanistic contributions of VAT and aberrant lipid metabolism to this process. The team includes clinical and translational researchers at two centers (UCSF and Duke) with expertise in NAFLD, PCOS, obesity, and lipid metabolism, with a track record of collaboration. The study team will leverage an existing well-characterized PCOS cohort29 to follow 150 reproductive-aged women with NASH (125 PCOS and 25 non-PCOS controls) to accomplish this.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic associated steatohepatitis (MASH) (formerly NASH)
* PCOS
* Non-PCOS

Exclusion Criteria:

* High levels of alcohol use (more than 7 drinks a week)
* Current pregnancy
* Other causes of hepatic steatosis
* Weight loss of more than 10% body weight in the last 6 months

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Our study population includes pre-menopausal women ages 18-42 years, 125 with PCOS and 25 non-PCOS controls, with probable or confirmed metabolic associated steatohepatitis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Liver Stiffness Change | from baseline to Year 3 follow- up.
  Mean change in liver stiffness (kPA) on magnetic resonance elastography (MRE)
Visceral Adipose Tissue (VAT) association to MASH severity | at baseline
  VAT volume (cm3) will be determined on magnetic resonance electrography (MRE)

SECONDARY OUTCOMES:
Liver stiffness severity | at baseline
  Severity of liver stiffness will be determined on magnetic resonance electrography (MRE)

CONTACTS AND LOCATIONS:
Overall Officials: Monika A Sarkar, M.D., M.A.S, Principal Investigator — University of California, San Francisco; Ayako Suzuki, M.D.,Ph.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No
At present all data collected will be de-identified and shared with only the researchers apart of this study.

REFERENCES:
- [Background] Sarkar M, Terrault N, Chan W, Cedars MI, Huddleston HG, Duwaerts CC, Balitzer D, Gill RM. Polycystic ovary syndrome (PCOS) is associated with NASH severity and advanced fibrosis. Liver Int. 2020 Feb;40(2):355-359. doi: 10.1111/liv.14279. Epub 2019 Nov 12. PMID 31627243
- [Background] Sarkar MA, Suzuki A, Abdelmalek MF, Yates KP, Wilson LA, Bass NM, Gill R, Cedars M, Terrault N; NASH Clinical Research Network. Testosterone is Associated With Nonalcoholic Steatohepatitis and Fibrosis in Premenopausal Women With NAFLD. Clin Gastroenterol Hepatol. 2021 Jun;19(6):1267-1274.e1. doi: 10.1016/j.cgh.2020.09.045. Epub 2020 Oct 1. PMID 33010412
- [Background] Sarkar M, Yates K, Suzuki A, Lavine J, Gill R, Ziegler T, Terrault N, Dhindsa S. Low Testosterone Is Associated With Nonalcoholic Steatohepatitis and Fibrosis Severity in Men. Clin Gastroenterol Hepatol. 2021 Feb;19(2):400-402.e2. doi: 10.1016/j.cgh.2019.11.053. Epub 2019 Dec 5. PMID 31812658
- [Background] Sarkar M, Terrault N, Duwaerts CC, Tien P, Cedars MI, Huddleston H. The Association of Hispanic Ethnicity with Nonalcoholic Fatty Liver Disease in Polycystic Ovary Syndrome. Curr Opin Gynecol Obstet. 2018 Feb 20;1(1):24-33. Epub 2018 Apr 5. PMID 30112518